CLINICAL TRIAL: NCT04151927
Title: Effects of an Overnight, 8-hour Low Oxygen Exposure on Resting Energy Expenditure and Appetite: a Pilot Study
Brief Title: Effects of Overnight Low Oxygen Exposure on Energy Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Claire E. Berryman, Assistant Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00000184
Record Dates: First submitted 2019-10-26; First posted 2019-11-05 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Resting Metabolic Rate; Appetite; Heart Rate Variability
Keywords: High altitude; Metabolic adaptations; Energy balance
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normobaric Hypoxia (NH) (Experimental): Overnight exposure (8 hours) to NH conditions (~15% oxygen; achieved with nitrogen dilution, equivalent to ~8500 feet elevation) using a commercially available tent and generator system (Hypoxico, Inc., New York, NY).
  Interventions: Device: Normobaric Hypoxia; Device: Normobaric Normoxia
- Normobaric Normoxia (NN) (Sham Comparator): Overnight exposure (8 hours) to NN conditions (~20% oxygen; achieved with nitrogen dilution, equivalent to ~1000 feet elevation) using a commercially available tent and generator system (Hypoxico, Inc., New York, NY).
  Interventions: Device: Normobaric Hypoxia; Device: Normobaric Normoxia

INTERVENTIONS:
Device: Normobaric Hypoxia — Low oxygen exposure to mimic ~8500 feet elevation.
Device: Normobaric Normoxia — Normal oxygen exposure to mimic ~1000 feet elevation (sham comparator).

SUMMARY:
This research study will evaluate changes in resting metabolic rate, appetite, and heart rate variability following overnight exposure (8 h/night) to normobaric hypoxia (NH) or normobaric normoxic (NN). In randomized order, participants will sleep one night in NH conditions (~15% oxygen; achieved with nitrogen dilution, equivalent to ~8500 feet elevation) and another night in NN (control) conditions (~20% oxygen; achieved with nitrogen dilution, equivalent to ~1000 feet elevation).

DETAILED DESCRIPTION:
Weight loss is a common factor reported in lowlanders traveling to high altitudes. Although the exact cause is unknown, studies have shown that weight loss at high altitude is associated with the amount of time and severity of the altitude exposure. Upon arrival to high altitude (≥ 5000 feet), numerous physiological adaptations occur that may promote weight loss, such as increased energy expenditure and reduced appetite. The breadth of current altitude research is limited by the logistical and monetary constraints of traveling to remote locations or access to an altitude chamber. A more logistically feasible alternative is the simulation of low oxygen conditions at sea level, using a commercially available tent and generator system to reduce ambient oxygen concentrations. The current research study will evaluate changes in resting metabolic rate, appetite, and heart rate variability following overnight exposure (8 h/night) to normobaric hypoxia (NH) or normobaric normoxic (NN). In randomized order, participants will sleep one night in NH conditions (~15% oxygen; achieved with nitrogen dilution, equivalent to ~8500 feet elevation) and another night in NN (control) conditions (~20% oxygen; achieved with nitrogen dilution, equivalent to ~1000 feet elevation). In the morning, following NH or NN exposure, resting metabolic rate will be measured using indirect calorimetry, appetite using an ad libitum buffet meal protocol, and heart rate variability by electrocardiogram. It is hypothesized that exposure to overnight NH will result in increased resting metabolic rate, decreased appetite, and decreased heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20 - 45 years
* Body mass index between 18.5 - 24.5 kg/m2
* Born at altitudes less than 2,100 meters (~7,000 feet)
* Currently residing in Tallahassee, Florida or the surrounding area
* Not taking any medication(s) that interfere with metabolism or oxygen delivery/transport for four weeks before and throughout the entire study (e.g., includes sedatives, sleeping aids, tranquilizers, and/or any medication that depresses ventilation, diuretics, alpha, and beta-blockers).
* Willing to refrain from smoking, vaping, chewing tobacco, and dietary supplement use throughout the entire study
* Willing to spend two overnight visits on the Florida State University campus.

Exclusion Criteria:

* Living in areas that are more than 1,200 m (~4,000 feet), or have traveled to areas that are more than 1,200 m for five days or more within the last two months
* Metabolic or cardiovascular abnormalities, gastrointestinal disorders, or any condition that interferes with metabolism or oxygen delivery/transport (e.g., kidney disease, diabetes, cardiovascular disease, etc.)
* Prior diagnosis of apnea or other sleeping disorders
* Prior diagnosis of high-altitude pulmonary edema or high-altitude cerebral edema
* Prior diagnosis of anemia or sickle cell anemia/trait
* Present condition of alcoholism, anabolic steroid, or other substance abuse issues
* Women who are pregnant, lactating, planning to become pregnant, or who have had an irregular menstrual cycle in the past six months.
* Allergies or intolerance to foods included in the standardized or ad libitum meal (e.g., lactose intolerance/milk allergy)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2021-10-02 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
Resting metabolic rate (kcal/d) following exposure to NH or NN conditions | 8 hours
  Resting metabolic rate will be accessed using indirect calorimetry (TrueOne 2400, Parvo Medics, Salt Lake City, UT) following 8 hours of overnight exposure to NH or NN.

SECONDARY OUTCOMES:
Objective appetite following exposure to NH or NN conditions | 8 hours
  Objective appetite will be assessed by measuring total energy intake during an ad libitum buffet-style meal provided to participants following 8 hours of overnight exposure to NH or NN.
Food preferences following exposure to NH or NN conditions | 8 hours
  Food preferences will be assessed by measuring macronutrient intake during an ad libitum buffet-style meal provided to participants following 8 hours of overnight exposure to NH or NN.
Fasting and postprandial hunger following exposure to NH or NN conditions | Hunger will be measured pre-meal (0 min), immediately post-meal, and at 15, 30, 45, 60, 90, and 120 min following 8 hours of NH or NN exposure
  Measures will be assessed before and after the ad-libitum buffet meal using visual analog scales following 8 hours of overnight exposure to NH or NN.
Fasting and postprandial satiety following exposure to NH or NN conditions | Satiety will be measured pre-meal (0 min), immediately post-meal, and at 15, 30, 45, 60, 90, and 120 min following 8 hours of NH or NN exposure
  Measures will be assessed before and after the ad-libitum buffet meal using visual analog scales following 8 hours of overnight exposure to NH or NN.
Fasting and postprandial prospective food consumption following exposure to NH or NN conditions | Prospective food consumption will be measured pre-meal (0 min), immediately post-meal, and at 15, 30, 45, 60, 90, and 120 min following 8 hours of NH or NN exposure
  Measures will be assessed before and after the ad-libitum buffet meal using visual analog scales following 8 hours of overnight exposure to NH or NN.
Fasting and postprandial subjective appetite following exposure to NH or NN conditions | Subjective appetite will be measured pre-meal (0 min), immediately post-meal, and at 15, 30, 45, 60, 90, and 120 min following 8 hours of NH or NN exposure
  Measures will be assessed before and after the ad-libitum buffet meal using visual analog scales following 8 hours of overnight exposure to NH or NN.
Energy intake following exposure to NH or NN conditions | 8 hours
  Energy intake will be accessed using the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool to complete dietary records for 2 days following 8 hours of overnight exposure to NH or NN.
Macronutrient intake following exposure to NH or NN conditions | 8 hours
  Macronutrient intake will be accessed using the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool to complete dietary records for 2 days following 8 hours of overnight exposure to NH or NN.
Heart rate variability following exposure to NH or NN conditions | 8 hours
  Heart rate variability will be measured using a 3-lead electrocardiogram following 8 hours of overnight exposure to NH or NN.
Prevalence of acute mountain sickness following exposure to NH or NN conditions | 8 hours
  Prevalence of acute mountain sickness will be accessed using the Environmental Symptoms Questionnaire following 8 hours of overnight exposure to NH or NN.
Severity of acute mountain sickness following exposure to NH or NN conditions | 8 hours
  Severity of acute mountain sickness will be accessed using the Environmental Symptoms Questionnaire following 8 hours of overnight exposure to NH or NN.
Continuous oxygen saturation during exposure to NH or NN | 8 hours
  Oxygen saturation will be measured continuously using a finger pulse oximeter (PalmSAT® 2500, Nonin Medical, Inc., Plymouth, MN) during 8 hours of overnight exposure to NH or NN.
Sleep quality following exposure to NH or NN conditions | 8 hours
  Sleep quality will be measured by the Pittsburgh Sleep Quality Index following 8 hours of overnight exposure to NH or NN.

CONTACTS AND LOCATIONS:
Overall Officials: Claire E Berryman, Ph.D., Principal Investigator — Department of Nutrition, Food, and Exercise Science at Florida State University.
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baker PA, Long AN, Dawson MA, Berryman CE. An Overnight, 8-Hour Low Oxygen Exposure Increases Energy Expenditure with No Effect on Energy Intake: A Randomized, Sham-Controlled, Crossover Study. J Nutr. 2026 Jan 5;156(3):101319. doi: 10.1016/j.tjnut.2025.101319. Online ahead of print. PMID 41500361